CLINICAL TRIAL: NCT02222402
Title: Evaluating the Clinical and Cost-effectiveness of Intra-dialytic Exercise for the Improvement of Health-related Quality of Life in People With Stage 5 Chronic Kidney Disease Undergoing Maintenance Haemodialysis Renal Replacement Therapy.
Brief Title: PrEscription of Intra-Dialytic Exercise to Improve quAlity of Life in Patients With Chronic Kidney Disease
Acronym: PEDAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIHR HTA Project Ref 12/23/09
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: End-Stage Kidney Disease
Keywords: Quality of Life; Exercise; Functional Capacity
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INTRA-DIALYTIC EXERCISE TRAINING (Experimental): Using a modified cycle ergometer, aerobic exercise will be performed in a semi-recumbent position, 3 times per week during the first two hours of haemodialysis. The initial prescription will be set in the moderate intensity range of 40-60% of peak aerobic capacity, progressing to 75% level by the end of the intervention.
  Twice per week patients will also complete lower extremity muscular conditioning exercise, using ankle weights, after the aerobic cycling exercise.
  Interventions: Behavioral: INTRA-DIALYTIC EXERCISE TRAINING
- HAEMODIALYSIS RENAL REPLACEMENT THERAPY (No Intervention): Haemodialysis is the most common dialysis (renal replacement) treatment for kidney failure.
  They may also receive dietary advice, counselling, input from social workers, and other forms of educational support.

INTERVENTIONS:
Behavioral: INTRA-DIALYTIC EXERCISE TRAINING
  Arms: INTRA-DIALYTIC EXERCISE TRAINING

SUMMARY:
The PEDAL study aims to evaluate the effectiveness of a 9-month intradialytic exercise training intervention designed to improve quality of life (QOL) and alleviate functional limitations in patients with stage 5 Chronic Kidney Disease (CKD) who are on haemodialysis. Exercise rehabilitation will be compared against established treatment options available within UK NHS haemodialysis (HD) units. A qualitative substudy will also investigate the experience and acceptability of the intervention for both participants and members of the renal care team. In addition, we want to examine whether this type of additional exercise treatment is cost effective within the health service setting.

PEDAL is designed as a multi centre randomised clinical trial (RCT) and will recruit 380 adult patients who have been on HD for at least 3 months, from 10 HD sites located in Scotland, England and Wales. The type of exercise programming will consist of cycling exercise performed during each dialysis session plus a muscle conditioning programme performed twice per week. All exercise sessions will be supervised by a physiotherapy assistant. The exercise prescription will be individualised for all patients on the basis of their fitness and clinical status.

The main objective is to examine the impact of exercise rehabilitation on quality of life and well being of patients. We hypothesise that the exercise training delivered during haemodialysis treatment will significantly improve the functional limitations/abilities of the patients leading to the detection of clinically beneficial improvement in quality of life outcome, as measured by the KDQOL-36 physical composite score (PCS) at the primary end point.

ELIGIBILITY:
Inclusion Criteria:

1. Prevalent Stage 5 CKD patients (GFR <15 mL/min) receiving maintenance haemodialysis therapy for more than 3 months
2. Male or female
3. Aged >18 years
4. Able to provide written informed consent

Exclusion Criteria:

1. Patients unlikely to be on HD for > 6 months - (this includes cachectic patients, those with severe heart failure, patients in whom dialysis withdrawal is being considered, and patients likely to receive a live-donor transplant or transfer to PD in that period of time);
2. Less than 3 months after the initiation of haemodialysis (patients in this time-frame are generally less clinically stable, many having vascular access procedures performed, and rates of inter-current events, including death and hospitalisation, are very much higher in the first 3 months after commencement of chronic haemodialysis);
3. Deemed to be clinically unstable by treating physician;
4. Dementia or severe cognitive impairment (as will be unable to give consent and/or complete questionnaire assessments);
5. Severe psychiatric disorders - except treated stable

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2015-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change from basline in quality of life on the Kidney Disease QOL questionnaire Physical Composite Score (KDQOL-PCS) at month 6. | Baseline, 6 months
  The KDQOL is a disease-specific quality of life measure.

CONTACTS AND LOCATIONS:
Overall Officials: Iain Macdougall, Study Chair — Kings College Hospital
Locations (1):
- Kings College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639